CLINICAL TRIAL: NCT06314321
Title: Baduanjin Exercise on Maintenance Hemodialysis Patients
Brief Title: The Effect of Baduanjin on Shoulder Function in Maintenance Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-K151-01
Record Dates: First submitted 2024-03-04; First posted 2024-03-18 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Hemodialysis Complication; Shoulder Joint Disorder; CKD-MBD
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin exercise group (Experimental): Before starting dialysis，Patients perform Baduanjin exercises. All Baduanjin training is provided by a professional doctor who has received training on BaduanJin and obtained certificate. Each session is approximately 30 minutes in duration, consisting of 5 minutes of warm-up exercises, 20 minutes of Baduanjinpractice, and 5 minutes of cool-down exercises.
  Interventions: Other: Baduanjin exercise
- Control group (No Intervention): Patients in this group maintain their conventional therapy and daily life activities, and there is no intervention given.

INTERVENTIONS:
Other: Baduanjin exercise — Baduanjin has 8 movement forms, which are relatively less demanding. Assistive equipment is also not necessary during Baduanjin. These advantages make Baduanjin a suitable form of exercise training for dialysis patients.The movements involved in Baduanjin require the individual to reach beyond the base of support, change the base of support between bilateral and unilateral stance, and perform movements in a sustained squatting posture. These maneuvers challenge balance and require muscle strength to be executed successfully. In 8 movement forms of Baduanjin all include shoulder joint function exercises, thus making Baduanjin a potentially useful method for improving activity level and arm strength.
  Arms: Baduanjin exercise group

SUMMARY:
The aim of this study is to examine the effect of 18-month Baduanjin exercise on shoulder joint function in maintenance hemodialysis (MHD) patients. 60 MHD patients aged 18-75 will included in this study and randomly divided into two groups (intervention group and control group). The intervention group will be led by a professional person and underwent Baduanjin exercise three times a week before hemodialysis. The control group maintained routine treatment and daily activities.

DETAILED DESCRIPTION:
The aim of this study is to observe the therapeutic effect of Baduanjin on improving shoulder joints in MHD patients. A total of 60 maintenance hemodialysis patients will be included and randomized into an intervention group of 30 cases and a control group of 30 cases. The intervention group underwent a 30 minute Baduanjin exercise under the guidance of a professional doctor before the dialysis day, including a 5-minute warm-up exercise, a 20 minute Baduanjin exercise, and a 5-minute relaxation exercise. The intervention group practice Baduanjin three days a week, while the control group maintain routine treatment and daily activities. Measure the indicators of each group at baseline, months 6, 12, and 18. The evaluation of shoulder joint function is based on the shoulder Constant score (which includes three dimensions: pain, daily living activities, and active range of motion); The quality of life score is based on the SF-12 score, and the emotional score is based on the Anxiety and Depression Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old, ≤ 75 years old
* Maintenance dialysis treatment for ≥ 3 months, three times a week
* The six minute walking experiment were used to screen patients for suitability for Baduanjin
* Right handedness, fistula in left hand

Exclusion Criteria:

* The vascular pathway is a tunnel catheter with a polyester sheath
* The vascular pathway is a right arteriovenous fistula
* Known infectious diseases
* Individuals with primary or secondary muscle diseases, mental abnormalities, lack of autonomous behavior ability, and lack of cooperation with clinical observation and treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Shoulder joint function score | 0 month，6 month，12 month，18 month
  Using the adjusted version of the CMS scoring scale, the total score is 75 points, including pain (15 points), daily living ability (ADL, 20 points), and joint range of motion (ROM, 40 points).
Shoulder joint internal rotation function | 0 month，6 month，12 month，18 month
  The patient takes a standing position and measures the distance between the fingers and vertebrae of the hemodialysis patient's fistulae and non fistulae hands, that is, the patient moves their thumb with the backhand as much as possible along the midline of the back, and uses a tape measure to measure the closest distance from the tip of their thumb to the spinous process of the 7th cervical vertebra. Relevant data is organized and recorded.
Muscle strength measurement | 0 month，6 month，12 month，18 month
  Grip strength can reflect the strength of the hand muscles, and a grip strength meter is used to measure the grip strength of the patient's hands separately. The patient takes a standing position, holds the handle with maximum force, and records the value when the number on the machine display screen no longer changes. Test three times, take the maximum value, and record the relevant results.
Area of biceps brachii muscle | 0 month，6 month，12 month，18 month
  Measure the thickness of the biceps brachii muscle in two groups of patients through skeletal muscle ultrasound examination.

SECONDARY OUTCOMES:
Changes in the Short Form-36 (SF-36) and European Quality of Life Five Dimension（EQ-5D-5L） | 0 month，6 month，12 month，18 month
  Changes from the Short Form-36 (SF-36) and European Quality of Life Five Dimension（EQ-5D-5L）scale at 0 months, 8 months, 12 months. The SF-12 score is used to evaluate an individual's health status and quality of life. The SF-12 score expressed as a number between 0 and 100, with higher numbers indicating better health. EQ-5D-5L evaluate quality of life from five aspects: action ability, self-care, daily activities, pain or discomfort, anxiety or depression. The score range generally ranges from less than 0 to 1, and the higher the score, the better the state; The VAS score range is 0-100, with higher scores indicating better health status.
Changes in the Hospital Anxiety and Depression Scale （HADS） | 0 month，6 month，12 month，18 month
  Changes from HADS Index at at 0 months, 8 months, 12 months. HADS consists of 14 items, of which 7 items assess depression and 7 items assess anxiety. The scores for anxiety and depression range from 0 to 21, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Li Yuan, MD, Study Chair — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Data can be shared after request

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT06314321/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT06314321/ICF_001.pdf